CLINICAL TRIAL: NCT06960395
Title: A Phase 1, First-in-Human Study of the Safety, Pharmacokinetics, and Preliminary Efficacy of VIR-5525 Alone and in Combination With Pembrolizumab in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: Safety and Preliminary Efficacy of VIR-5525 and VIR-5525 + Pembrolizumab in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIR-5525-V101; U1111-1294-8156 (Registry Identifier: ICTRP); 2023-508555-39 (Registry Identifier: CTIS); AMX-525 (Other: Amunix)
Record Dates: First submitted 2025-04-21; First posted 2025-05-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor Malignancies; EGFR Positive Solid Tumors; EGFR
Keywords: VIR-5525
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: VIR-5525 Monotherapy Dose Escalation (Experimental): Screening Period: Up to 28 days
  Treatment Period: Once successfully screened, enrolled participants may receive study intervention of VIR-5525 in monotherapy.
  Interventions: Drug: VIR-5525
- Part 2: VIR-5525 Monotherapy Dose Expansion (Experimental): Screening Period: Up to 28 days
  Treatment Period: Once successfully screened, enrolled participants may receive study intervention of VIR-5525 in monotherapy.
  Interventions: Drug: VIR-5525
- Part 3: VIR-5525 Combination Dose Escalation (Experimental): Screening Period: Up to 28 days
  Treatment Period: Once successfully screened, enrolled participants may receive study intervention of VIR-5525 in combination with pembrolizumab.
  Interventions: Drug: VIR-5525; Drug: Pembrolizumab
- Part 4: VIR-5525 Combination Dose Expansion (Experimental): Screening Period: Up to 28 days
  Treatment Period: Once successfully screened, enrolled participants may receive study intervention of VIR-5525 in combination with pembrolizumab.
  Interventions: Drug: VIR-5525; Drug: Pembrolizumab

INTERVENTIONS:
Drug: VIR-5525 — Pharmaceutical Form: Solution for Infusion Route of Administration: Intravenous (IV) infusion
  Other Names: AMX-525
Drug: Pembrolizumab — Pharmaceutical Form: Solution for Infusion Route of Administration: Intravenous (IV) infusion
  Arms: Part 3: VIR-5525 Combination Dose Escalation; Part 4: VIR-5525 Combination Dose Expansion

SUMMARY:
This Phase 1, first-in-human (FIH), dose-escalation and dose-expansion study is designed to evaluate the safety, PK, and preliminary anti-tumor activity of VIR-5525 as a monotherapy and in combination with pembrolizumab in participants with solid tumors that are known to express EGFR.

The study will be conducted in the following 4 parts:

* Part 1: VIR-5525 monotherapy dose escalation
* Part 2: VIR-5525 monotherapy dose expansion
* Part 3: VIR-5525 plus pembrolizumab dose escalation
* Part 4: VIR-5525 plus pembrolizumab dose expansion

ELIGIBILITY:
Inclusion Criteria:

I 01. Are ≥ 18 years of age, or at the country's legal age of majority of the legal adult age is >18 years, at the time of signing the ICF.

I 02. Have an ECOG performance status of 0 to 1.

I 03. Have a life expectancy of at least 12 weeks.

I 04. Have histological, pathological, or cytological confirmation of disease type that is unresectable, locally advanced, or metastatic.

I 05. Have measurable disease per RECIST v1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

I 06. Have diseases under study, lines of therapy, and biomarker status, as follows:

Have one of the following:

• (Parts 1 and 3): NSCLC (nonsquamous or squamous histology), CRC, HNSCC, or CSCC.

Note: Participants with nasopharyngeal tumors are eligible. Note: Participants with upper esophageal or salivary gland tumors are not eligible.

OR

• Have a solid tumor with EGFR amplification (as previously determined locally with an analytically validated assay in a certified testing laboratory).

Have no available standard systemic therapy; or standard therapy is intolerable, not effective, or not accessible; or participant has refused standard therapy.

Exclusion Criteria:

E 01. Are a WOCBP with a positive serum or urine pregnancy test within 72 hours prior to treatment.

E 02. Have acute or chronic infections, including the following:

* Acute or chronic active Epstein-Barr virus (EBV) infection (Exception: asymptomatic EBV-positive participants are still eligible)
* Chronic active EBV disease defined as a chronic illness lasting at least 6 months, an increased EBV level in either the tissue or the blood, and lack of evidence of a known underlying immunodeficiency
* History of hepatitis B infection (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) infection (defined as HCV [HCV RNA; qualitative] is detected)
* History of HIV infection. No HIV testing is required unless mandated by the local health authority.
* Active infection requiring systemic therapy within 14 days of Cycle 1 Day 1
* Known positive COVID-19 test result at screening (Exception: If follow-up test is negative, participants may be eligible if asymptomatic and upon consultation with medical monitor)

E 03. Have a concomitant medical or inflammatory condition that may increase the risk of toxicity to VIR-5525 or pembrolizumab, per the investigator

E 04. Have a QT interval corrected by Fridericia's method (QTcF) that is >480 ms

E 05. Have received prior systemic anti-cancer therapy, including investigational agents, within 5 half-lives prior to first dose of study intervention. For drugs with a long t1/2, such as mAbs, or for drugs for which the t1/2 is not known, the last dose should not have been within 28 days prior to first dose of study intervention.

Note: If the participant has had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.

E 06. Have received prior radiotherapy within 2 weeks of start of study intervention Note: Participants must have recovered from all radiation-related toxicities to Grade ≤1 or baseline, must not require corticosteroids, and must not have had radiation pneumonitis.

Exception: External beam radiotherapy, including palliative external radiation, is allowed.

A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Objectives (Parts 1 and 3) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To evaluate the safety and tolerability of escalating doses of VIR-5525 as monotherapy (Part 1) and in combination with pembrolizumab (Part 3).
  Endpoint: Incidence and severity of AEs, including DLTs, with severity determined according to NCI CTCAE v5.0, ASTCT CRS, or ASTCT ICANS Consensus Grading, as appropriate.
Primary Safety Objectives (Parts 1 and 3) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To determine the recommended dose(s) for expansion cohorts of VIR-5525 as monotherapy (Part 1) and in combination with pembrolizumab (Part 3).
  Endpoint: Incidence and severity of AEs, including DLTs, with severity determined according to NCI CTCAE v5.0, ASTCT CRS, or ASTCT ICANS Consensus Grading, as appropriate.
Primary Efficacy Objectives (Parts 2 and 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To evaluate the preliminary anti-tumor activity of VIR-5525 as monotherapy (Part 2) and in combination with pembrolizumab (Part 4) at the recommended dose(s) for expansion cohorts.
  Endpoint: Objective response, defined as a CR or PR per RECIST v1.1.

SECONDARY OUTCOMES:
Secondary Safety Objectives (Parts 1 and 3) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To further evaluate the safety and tolerability of VIR-5525 as a monotherapy (Part 2) and in combination with pembrolizumab (Part 4).
  Endpoint: Incidence and severity of AEs, with severity determined according to NCI CTCAE v5.0, ASTCT CRS, or ASTCT ICANS Consensus Grading, as appropriate.
Secondary Efficacy Objectives (Parts 1 and 3) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To evaluate the preliminary anti-tumor activity of VIR-5525 as monotherapy (Part 1) and in combination with pembrolizumab (Part 3).
  Endpoint: Objective response, defined as a CR or PR per RECIST v1.1.
  Endpoint: DOR, defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs first, per RECIST v1.1.
Secondary Efficacy Objectives (Parts 2 and 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To further evaluate the preliminary anti-tumor activity of VIR-5525 as monotherapy (Part 2) and in combination with pembrolizumab (Part 4) at the recommended dose(s) for expansion cohorts and schedule.
  Endpoint: DOR, defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs first, per RECIST v1.1.
Secondary Efficacy Objectives (Parts 2 and 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To further evaluate the preliminary anti-tumor activity of VIR-5525 as monotherapy (Part 2) and in combination with pembrolizumab (Part 4) at the recommended dose(s) for expansion cohorts and schedule.
  Endpoint: PFS (per investigator using RECIST v1.1), defined as the length of time from the start of treatment until first documented disease progression or death.
Secondary PK Objectives (Parts 1 Through 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To characterize the PK profile of VIR-5525 as monotherapy (Parts 1 and 2) and in combination with pembrolizumab (Parts 3 and 4).
  Endpoint: PK parameters of VIR-5525, including, but not limited to, area under the curve (AUC), calculated as data allow.
Secondary PK Objectives (Parts 1 Through 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To characterize the PK profile of VIR-5525 as monotherapy (Parts 1 and 2) and in combination with pembrolizumab (Parts 3 and 4).
  Endpoint: PK parameters of VIR-5525, including, but not limited to, maximum concentration of the drug (Cmax), calculated as data allow.
Secondary PK Objectives (Parts 1 Through 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To characterize the PK profile of VIR-5525 as monotherapy (Parts 1 and 2) and in combination with pembrolizumab (Parts 3 and 4).
  Endpoint: PK parameters of VIR-5525, including, but not limited to, time to peak drug concentration (tmax), calculated as data allow.
Secondary PK Objectives (Parts 1 Through 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To characterize the PK profile of VIR-5525 as monotherapy (Parts 1 and 2) and in combination with pembrolizumab (Parts 3 and 4).
  Endpoint: PK parameters of VIR-5525, including, but not limited to, drug accumulation ratio (Rac), calculated as data allow.
Secondary Immunogenicity Objectives (Parts 1 Through 4) | From Cycle 1, Day 1 (each cycle is 21 days), up to approximately 52 months.
  Objective: To evaluate the immunogenicity of VIR-5525 as monotherapy (Parts 1 and 2) and in combination with pembrolizumab (Parts 3 and 4).
  Endpoint: Incidence of ADAs to VIR-5525 at baseline and incidence of treatment-emergent ADAs to VIR-5525.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Vir Biotechnology
Locations (3):
- Honor Health Research Institute, Scottsdale, Arizona, United States
- Australia (2):
  - Wollongong Hospital, Wollongong, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland

IPD SHARING:
Plan to Share IPD: No